CLINICAL TRIAL: NCT01554384
Title: Multicentre Randomised Control Trial of Point-of-treatment (Clinic-based) Xpert MTB/RIF Assay
Brief Title: Trial of Point-of-treatment Xpert MTB/RIF Assay
Acronym: TBNEATXpert
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Biomedical Research and Training Institute (Other); University of Zimbabwe (Other); University of Zambia (Other); Medical Research Council, South Africa (Other); Mbeya medical research program (Unknown); McGill University (Other); Radboud University Medical Center (Other); University of Cape Town Lung Institute (Other)
Responsible Party: Principal Investigator, Keertan Dheda, Professor and Head, Lung Infection and Immunity unit, University of Cape Town
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: TBNEATXpertRCT; IP.09.32040.009 (Other Grant/Funding Number: EDCTP)
Record Dates: First submitted 2011-07-07; First posted 2012-03-15 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; diagnosis; Xpert MTB/RIF; point-of-treatment; randomized controlled trial
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xpert MTB/RIF (Experimental): Patients in this arm will receive 1 sputum Xpert MTB/RIF test (point-of-treatment) and 1 sputum sample for MGIT liquid TB culture (regional lab)
  Interventions: Procedure: Xpert MTB/RIF assay
- Sputum smear microscopy (Active Comparator): Patients in this study arm will receive 2 sputum samples for same-day smear microscopy and 1 of the sputum samples will have a MGIT Liquid culture (regional lab).
  Interventions: Procedure: Smear microscopy

INTERVENTIONS:
Procedure: Xpert MTB/RIF assay — Automated nucleic-acid amplification test (fully integrated) test for TB
  Other Names: Cepheid Xpert MTB/RIF assay
  Arms: Xpert MTB/RIF
Procedure: Smear microscopy — Smear microscopy involve sputum smear with either ziehl-neelsen or auramine-O staining of slides and light or fluorescence microscopy reading
  Arms: Sputum smear microscopy

SUMMARY:
Xpert MTB/RIF assay is a novel automated molecular tool for the diagnosis of TB. Xpert can detect TB genetic material in sputum samples as well as test for genetic resistance to rifampicin providing results within 2 hours. Xpert received WHO endorsement in December 2010. There is limited data on the impact of Xpert on time-to-treatment and TB-related patient morbidity in primary care clinics. No studies have yet evaluated Xpert performed at the point-of-treatment (POT) i.e. in primary care clinic location. The investigators hypothesize that one sputum GeneXpert MTB/RIF assay performed at the POT will improve time-to-diagnosis, time-to-treatment and TB related patient morbidity for patients with suspected TB presenting to primary level TB clinics in high HIV prevalent settings.

DETAILED DESCRIPTION:
Tuberculosis (TB) is one of the world's most important infectious causes of mortality and continues to kill 1.8 million people annually. Despite intensified standard measure of TB control, TB case detection rates are low, posing major hurdles for TB control. It is estimated that approximately 50% of patients with TB are still not diagnosed and treated appropriately. The problem is compounded by the increasing prevalence of multi drug resistant (MDR) and extensively drug resistant (XDR) TB and the close association between TB and HIV infection.

Diagnostic tools introduced 100 years ago are still in routine use and increasingly inaccurate if the face of the HIV and TB syndemics. Consequently, many patients with active TB remain undiagnosed and continue to spread the disease within the community. Thus, missed or delayed diagnosis results in ongoing transmission, patient morbidity and mortality, and social and economic consequences. Currently, there is no available point-of-care, or even point-of-treatment test that allows early detection of active tuberculosis at the peripheral health clinic level. Lack of rapid, simple and accurate diagnostic tests at this level is a major hurdle in controlling the global burden of TB. A number of promising new TB diagnostics have shown initial promise but there remains an urgent need to assess their impact when used at the point-of-treatment in primary care level.

In 2009, Cepheid released the Xpert® MTB/RIF Assay, which is the only system able to deliver answers directly from unprocessed samples by combining on-board preparation of the sample with real-time polymerase chain reaction (PCR) in less than 2 hours. Additionally, the Xpert® MTB/RIF Assay allows for simultaneous on-demand molecular testing for the detection of mycobacterium tuberculosis (M.tb) and rifampicin (frontline anti-TB drug) resistance. . The GeneXpert™ system consists of a GeneXpert instrument, personal computer and disposable fluidic cartridges. The system combines cartridge-based sample preparation with amplification and detection in a fully integrated and automated nucleic acid analysis instrument. Xpert has now been shown to be an accurate tool for the rapid diagnosis of tuberculosis in both smear-positive and smear-negative samples in both a multicentre evaluation and demonstration study with a sensitivity of approximately 70% in smear negative culture positive TB. Xpert testing in both these studies was performed at microscopy laboratories. In December 2010, on the basis of these results, Xpert was endorsed for TB diagnosis by the World Health Organisation (WHO) but is yet to be integrated into national tuberculosis control programmes.

Limited data is available on the impacts of Xpert on patient important outcomes such as TB-related morbidity. No data is available about the feasibility and robustness of performing Xpert in primary care clinics at the POT using minimally trained nursing staff. The objective of this study will be to examine the feasibility and impact of a single point-of-treatment Gene Xpert MTB/RIF Assay performed by clinic staff compared to standard microscopy-centre based diagnostics. Special focus will be on the patient-related outcomes of time-to-treatment initiation, drop out rates and the mean difference in TB-morbidity scores in patients diagnosed with Xpert.

The Xpert POT study will be a multicentre patient-level randomised controlled trial comparing a single sputum GeneXpert MTB/RIF Assay performed at point-of-treatment with same-day standard fluorescent smear microscopy for TB diagnosis at the primary level of care. A single liquid MGIT culture performed a regional laboratory will be used as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give informed consent
2. Ambulant patient presenting to TB clinic

   IF HIV negative requires 2 or more of the following:
   * Cough ≥ 2 weeks
   * loss of weight
   * persistent fever ≥ 2 weeks and/or
   * a single recorded temp > 38°C
   * night sweats
   * generalized fatigue
   * hemoptysis or
   * chest pain

   OR if HIV positive - any one of the following:
   * current cough
   * night sweats
   * fever
   * loss of weight
3. Patient 18 years or above

Exclusion Criteria:

1. Inability to provide informed consent (e.g. mentally impaired)
2. Unable to produce 2 sputa of ≥ 1ml
3. TB treatment within the last 60 days
4. Unable to potentially return for study follow-up at 2 and 6 months (i.e. leaving community)
5. Patient not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1472 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Difference in TB-related Morbidity | 2 months
  Time-specific (2 month) difference in morbidity between the Xpert MTB/RIF and smear microscopy study arms.
  Morbidity will be assessed using the TB Score and Karnosky performance scale
Difference in TB-related Morbidity | 6 months
  Time-specific (6 month) difference in morbidity between the Xpert MTB/RIF and smear microscopy study arms.
  Morbidity will be assessed using the TB Score and Karnosky performance scale

SECONDARY OUTCOMES:
Time-to-diagnosis | 6 months
  Time from study enrollment to TB diagnosis in each study arm
  A diagnosis of TB will include:
  i) Smear microscopy: WHO classification for smear grading considered positive ii) Xpert MTB/RIF positive (mtb detected) iii) MGIT liquid culture positive
Drop-out and lost-to-follow up rates | 1 year
  Number of patients that are enrolled, randomized to a study arm, and then do not return to receive a positive test result, and Number of patients that are enrolled, randomized to a study arm, diagnosed with TB, and then are lost-to-follow up prior to completion of prescribed standard TB treatment
Feasibility of clinic-based performance of Xpert MTB/RIF assay performed by nursing staff without formal research training | 6 months
  Feasibility indicators for the performance of Xpert at POT will be recorded. These include indeterminate rates, turn-around-time, user appraisal and assessments and performance comparisons between laboratory and clinic-based Xpert MTB/RIF.
Individual patient-level cost analysis, cost-effectiveness evaluation and quality of health indices evaluation | 1 year
  Detailed documentation of patient and health system costs for TB diagnosis and treatment will be done at baseline, 2 month and 6 month time-points as well as quality of life health questionaires.
Time-to-treatment initiation | 6 months
  The time-to-treatment initiation for TB culture positive patients in each study arm will be compared Treatment commencement will be considered as the initiation of the first dose of anti-TB treatment at a registered DOTs facility

CONTACTS AND LOCATIONS:
Overall Officials: Keertan Dheda, MD PhD, Principal Investigator — University of Cape Town
Locations (4):
- South Africa (2):
  - Medical Research Council, Durban, KwaZulu-Natal
  - University of Cape Town, Cape Town, Western Cape
- University Teaching Hospital of Zambia, Lusaka, Zambia
- University of Zimbabwe, Harare, Zimbabwe

REFERENCES:
- [Derived] Theron G, Zijenah L, Chanda D, Clowes P, Rachow A, Lesosky M, Bara W, Mungofa S, Pai M, Hoelscher M, Dowdy D, Pym A, Mwaba P, Mason P, Peter J, Dheda K; TB-NEAT team. Feasibility, accuracy, and clinical effect of point-of-care Xpert MTB/RIF testing for tuberculosis in primary-care settings in Africa: a multicentre, randomised, controlled trial. Lancet. 2014 Feb 1;383(9915):424-35. doi: 10.1016/S0140-6736(13)62073-5. Epub 2013 Oct 28. PMID 24176144